CLINICAL TRIAL: NCT05537311
Title: Reducing Isolation and Loneliness in Patients With Critical Illness With Novel Engagement Strategies: a Pilot Randomized Trial
Brief Title: Reducing Isolation and Feeling of Loneliness During Critical Illness
Acronym: SOCIAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kirby Mayer (Other)
Responsible Party: Sponsor-Investigator, Kirby Mayer, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 77702
Record Dates: First submitted 2022-07-27; First posted 2022-09-13 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Critical Illness; Social Isolation; Anxiety; Depression; Post Intensive Care Unit Syndrome
Keywords: critical illness; Post Intensive Care Unit Syndrome; social isolation
MeSH Terms: conditions — Critical Illness; Social Isolation; Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: pilot-randomized trial
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor will be blinded to treatment group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Social engagement using VR (Experimental): Patients will receive social engagement with emphasize on meaningful conversation, cognitive engagement, and emotional support provided by trained research assistant using virtual reality as a vehicle for delivery. Subjects will receive 15-45 minutes of treatment per day for 5 days initiated after respiratory support (Intubation via mask or tube, high-flow nasal cannula) have been weaned to nasal cannula. Experimental group will also receive standard of care
  Interventions: Behavioral: Social Engagement
- Control (No Intervention): Control will receive standard of care

INTERVENTIONS:
Behavioral: Social Engagement — 30-45 minutes of social engagement provided to patients in ICU. Social engagement strategies including meaningful conversation, cognitive stimulation, and emotional support
  Arms: Social engagement using VR

SUMMARY:
The trial is a pilot-randomized trial testing feasibility and limited-efficacy of delivering social engagement using technologic strategies to reduce periods of social isolation.

DETAILED DESCRIPTION:
Patients with critical illnesses such as sepsis and acute respiratory failure (ARF) who require an ICU stay are at high risk of developing anxiety, depression, post-traumatic stress disorder, and cognitive deficits. Risk factors for emotional and cognitive impairments after ICU include underlying systematic illness, as well as consequences of life-saving therapies. In brief, patients are frequently restricted and even restrained to the bed, provided high dosages of sedatives, develop delirium, and are isolated from family and staff for extended periods of time. Moreover, the ICU environment including lights, noises, and the social isolation have a serious negative impact on cognitive function and emotional health status. Prospective data from the ICU demonstrate that critically ill patients in ICU spend two-thirds of their time completely alone.

Patients who have survived describe their ICU experience as a traumatic event similar to war, and testimonials for the ICU Recovery clinic frequently resemble: "I felt like I was being held captive in an unknown basement." Periods of social isolation in daily life as well as in the hospital have a significant negative impact on patient-centered outcomes including increased risk of disability, frailty, and mortality. Our study will examine the feasibility of delivering social engagement interventions using technology such as virtual reality (VR) to reduce feelings of isolation and loneliness. There have been a handful of projects to reduce anxiety and depression using a myriad of delivery techniques including journaling in a diary, emotional-behavioral therapy, face-to-face social engagement and family engagement using face-time and VR. These projects, however, have not examined the impact of social engagement on reducing periods of isolation and loneliness. We hypothesize that social engagement delivered using VR technologies will reduce periods of social isolation and thus improve anxiety, depression, and post-traumatic stress disorder (PTSD).

ELIGIBILITY:
Inclusion Criteria:

* adult
* admitted to ICU with acute respiratory failure (ventilation via tube or mask or HFNC)

Exclusion Criteria:

* previous cognitive or emotional health condition
* inability to follow commands

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2022-07-27 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Feasibility of implementing the study intervention | Through completion of the intervention, which on average will occur one week after randomization
  Determine the number of sessions delivered per number of sessions scheduled. The study sample size of 12 subjects to receive the intervention, and each subject in the intervention should receive 5 sessions each = 60 sessions total; success will be considered 75% of sessions delivered (45 sessions completed of 60 planned).
Safety of the study intervention defined as number of patients with treatment-related adverse event | Through completion of the intervention, which on average will occur one week after randomization
  Minor adverse events, major adverse events, and unanticipated problems as assessed by the investigators per study protocol will be recorded during each treatment session. The rate of adverse events will be examined.

SECONDARY OUTCOMES:
Self-reported anxiety | Through study completion, which will occur on average 1-3 months after hospital discharge
  Hospital Anxiety and Depression Scale - Anxiety- self report questionnaire with higher scores indicating worse perceived anxiety
Self-reported depression | Through study completion, which will occur on average 1-3 months after hospital discharge
  Hospital Anxiety and Depression Scale - Depression - self report questionnaire with higher scores indicating worse perceived depression
Self-reported health related quality of life | Through study completion, which will occur on average 1-3 months after hospital discharge
  EurQol-5Domain (EQ-5D) - self report questionnaire with higher scores indicating better perceived quality of life
Cognitive function | Through study completion, which will occur on average 1-3 months after hospital discharge
  Montreal Cognitive Assessment - performed cognitive examination with higher scores indicating better cognitive function

CONTACTS AND LOCATIONS:
Locations (1):
- UK Heatlhcare, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Undecided
IPD will be shared via dissemination at national conferences and manuscripts; and available upon request of the primary investigator